CLINICAL TRIAL: NCT00951587
Title: Evaluation of the PillCam™ Colon Capsule Endoscopy (PCCE) Night Procedure
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Corporate Manager Clinical Affiars, Given Imaging Ltd.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MA-104
Record Dates: First submitted 2009-08-02; First posted 2009-08-04 (Estimated); Last update posted 2019-07-31 (Actual); Status verified 2010-03

CONDITIONS: Colonic Diseases
Keywords: Colonic Diseases
MeSH Terms: conditions — Colonic Diseases | interventions — Capsule Endoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Patients that are indicated for colonoscopy or who are suspected or known to suffer from colonic diseases.
  Interventions: Device: PillCam™ (Capsule Endoscopy)

INTERVENTIONS:
Device: PillCam™ (Capsule Endoscopy) — Medical Device

SUMMARY:
The purpose of this study is to evaluate the effect of the night procedure in regards to colon cleansing level and capsule excretion rate.

DETAILED DESCRIPTION:
The evaluation of subjects with suspected colonic disease includes endoscopic imaging by colonoscopy and radiologic imaging such as air-contrast barium enema, or CT colonography. The Given® Diagnostic System offers an alternative approach for endoscopic visualization of the colon using capsule endoscopy, an ingestible device which contains imagers, light sources, a power source and a RF transmitter. Advantages of the Given® Diagnostic System include the elimination of the need for sedation, the minimally invasive, painless nature of the exam, and the ability to pursue normal daily activities immediately following the procedure . Furthermore, compared to standard colonoscopy, the Given® Diagnostic System may be more readily accepted by the subjects, thereby improving subjects' willingness to undergo a diagnostic evaluation of the colon and comply with colorectal cancer screening recommendations.

The PillCam™ SB capsule (formerly M2A® Capsule) that was FDA-approved in August 2001 for small bowel evaluation has been ingested to date by more than 500,000 people worldwide and is well accepted by patients and physicians as well as the processional societies. However, adequate visualization of the colon cannot be achieved with the standard PillCam™ SB capsule because of the anatomical and physiological properties of the colon which are significantly different than the small bowel. Moreover, other issues that limit the evaluation of the colonic mucosa by the standard PillCam™ SB procedure include an unsatisfactory level of colon cleanliness and slow progression of the PillCam™ SB capsule through the colon during the desired examination time. Therefore, the development and introduction of a specially designed, customized colon capsule combined with a dedicated capsule colonoscopy procedure protocol will allow for more efficient evaluation of the colonic mucosa. This is expected to improve the capability of the Given® Diagnostic System to detect colonic pathologies and to serve as a diagnostic and screening tool for colonic disease. Further details of the PillCam™ Colon Capsule Endoscope (PCCE) can be found in the device description section.

This is a pilot study that is designed to evaluate the level of cleanliness and visualization of colon achieved by colon capsule endoscopy when using Night procedure regimens for preparation of the colon.

ELIGIBILITY:
Inclusion criteria:

* Subject is between the ages of 50-75 years and has an indication to undergo colonoscopy: At least 75% of total cases OR
* Subject is 18-50 suspected/known to suffer from large bowel disease and was clinically referred for colonoscopy (e.g. rectal bleeding, melena, positive FOBT, recent change of bowel habits, CRC screening, UC, positive findings on a GI radiographic study - no more than 25% of total cases

Exclusion criteria

* Subject has dysphagia or any swallowing disorder
* Subject has severe Congestive heart failure (NYHA II or IV)
* Subject has renal insufficiency
* Subject has had prior abdominal surgery of the gastrointestinal tract other than uncomplicated procedures that would be unlikely to lead to bowel obstruction based on the clinical judgement of the investigator
* Subject has a cardiac pacemaker or other implanted electromedical device.
* Subject has any allergy or other known contraindication to the medications used in the study
* Subject is expected to undergo MRI examination within 7 days after ingestion of the capsule.
* Subject with any condition believed to have an increased risk for capsule retention such as Crohn's disease, intestinal tumors, radiation enteritis, or NSAID enteropathy,
* Subject has any condition, which precludes compliance with study and/or device instructions.
* Women who are either pregnant or nursing at the time of screening, who intend to be during the study period, or are of child-bearing potential and do not practice medically acceptable methods of contraception.
* Subject suffers from life threatening conditions
* Subject currently participating in another clinical study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2008-02; Primary Completion 2010-02 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Colon cleansing level score | within 7 days
Transit time in the different GI regions until excretion | within 7 days

SECONDARY OUTCOMES:
Accuracy parameters of PCCE, compared to colonoscopy | within 7 days
Number of complete capsule procedure | within 7 days
Patient subjective assessment questionnaires | within 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Wolff Schmiegel, Prof. Dr., Principal Investigator — Knappschaftskrankenhaus Medizinische Universitaetsklinik
Locations (2):
- Germany (2):
  - Berufsgenossenschaftliche Universitätskliniken Bergmannsheil, Bochum
  - Knappschaftskrankenhaus Medizinische Universitaetsklinik, Bochum